CLINICAL TRIAL: NCT06533267
Title: Endoscopic Surgery Compared With Intensity Modulated Radiotherapy for Stage I Nasopharyngeal Carcinoma : A Multicenter, Randomized Controlled Clinical Trial.
Brief Title: Endoscopic Surgery vs. Intensity Modulated Radiotherapy for Stage I Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Huazhong University of Science and Technology Union ShenZhen Hospital (Nanshan Hospital) (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professior, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2024-02-24
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma; Intensity Modulated Radiotherapy; Surgery
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery plus close follow-up (Experimental): Surgery:
  Endoscopic Nasopharyngectomy: Radical resection of the primary lesion using nasal endoscopy.
  Interventions: Procedure: Endoscopic nasopharyngectomy followed close follow-up
- Intensity modulated radiotherapy (Active Comparator): Radiotherapy:
  Intensity-modulated Radiotherapy:
  GTVnx: 69.96Gy/33Fr/2.12Gy CTV1: 59.4Gy/33Fr/1.8Gy CTV2: 54.12Gy/33Fr/1.64Gy
  Interventions: Radiation: Intensity-modulated Radiotherapy

INTERVENTIONS:
Procedure: Endoscopic nasopharyngectomy followed close follow-up — Radical resection of primary lesion using nasal endoscopy.
  After the treatment, the electronic nasal endoscopy was reviewed every two weeks to determine the healing of the wound, whether there was tumor recurrence, until the surgical wound was completely healed. The patients were followed up at least once every three months from the first year to the third year, at least once every six months from the fourth year to the fifth year, and at least once every year after five years.
  Arms: Surgery plus close follow-up
Radiation: Intensity-modulated Radiotherapy — GTVnx (nasopharyngeal lesions): 69.96Gy/33Fr/2.12Gy CTV1: 60.60Gy/33Fr/1.82Gy CTV2: 54.12Gy/33Fr/1.64Gy.
  After treatment, patients were followed up every 3-6 months from the first year to the third year, every 6-12 months from the fourth year to the fifth year, and at least once a year after five years.
  Arms: Intensity modulated radiotherapy

SUMMARY:
The goal of this clinical trial is to compare the survival and adverse reactions differences between endoscopic surgery and intensity modulated radiotherapy for patients with newly diagnosed stage Ⅰ nasopharyngeal carcinoma, aiming to verifying the efficacy and safety of endoscopic surgery for stage Ⅰ nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
The newly diagnosed non-metastatic nasopharyngeal carcinoma has shown satisfactory therapeutic effect under the intensity modulated radiation. The 5-year survival rate of the newly diagnosed Ⅰ nasopharyngeal carcinoma was more than 95%. However, mos patients receiving radical radiotherapy will experience different degrees of acute or chronic radiation injury, which will affect the quality of life of patients to varying degrees. For stage Ⅰ nasopharyngeal carcinoma with primary lesion confined to nasopharyngeal mucosa and without regional lymph node metastasis, in theory, the primary lesion can be removed by minimally invasive surgery without need of preventive treatment of cervical lymph nodes according to the prior study.

Based on our previous research results, we stratified the nasopharyngeal primary tumor diameter of stage Ⅰ nasopharyngeal carcinoma by whether the short diameter of retropharyngeal lymph nodes and neck lymph nodes was smaller than 0.4cm and 0.6cm respectively, and the tumor diameter of nasopharyngeal primary tumor was ≤ 1.5cm. This study evaluated the efficacy and safety of endoscopic minimally invasive surgery compared to conventional intensity-modulated radiotherapy for these stage Ⅰ nasopharyngeal carcinoma.

In this study, the stage Ⅰ patients in the experimental group only received endoscopic nasopharynx resection and were followed up closely to monitor the recurrence and distant metastasis of the tumor.

The patients in the control group received conventional intensity-modulated radiotherapy and regular follow-up. The target area and dose of radiotherapy were as follows: GTVnx: primary lesion of the nasopharynx; CTV1: high-risk area and the entire nasopharynx; CTV2: low-risk area. The recommended intensity-modulated radiotherapy dose is GTVnx(69.96 Gy/33 Fr/2.12 Gy); CTV1(60.60 Gy/33 Fr/1.82 Gy); CTV2(54.12 Gy/33 Fr/1.64 Gy).

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky score >70.
* Non-keratinized carcinoma of the nasopharynx (differentiated or undifferentiated, i.e., WHO type II or III) or carcinoma in situ confirmed histologically and/or cytologically.
* According to the eighth edition of UICC/AJCC staging, the patient was defined as T1N0M0 stage I.
* The maximum short diameters of retropharyngeal lymph nodes and cervical lymph nodes were not more than 0.4cm and 0.6cm respectively, or retropharyngeal lymph nodes and cervical lymph nodes were 0.4-0.5cm and 0.6-1.0cm respectively but PET/CT showed negative.
* Informed Concent signed with willingness to obey the follow-up, treatment, examination and any other programs according to the research protocol.

Exclusion Criteria:

* MRI showed that the primary tumor diameter >1.5cm, or internal carotid artery vascular malformation which would seriously affect the operation.
* Diagnosed as recurrent or distant metastatic nasopharyngeal carcinoma or together with any other malignancy.
* Suffering severe organ dysfunction or physical disorder which could not tolerate operation or radiotherapy.
* Unable to cooperate with regular follow-up due to psychological, social, domestic or geological reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2034-03-25 (Estimated); Study Completion 2034-03-25 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Defined as the time interval from randomization to death due to any cause.
Incidence of ≥3 grade adverse events | 5 years
  The proportion of patients with ≥3 grade adverse events according to CTCAE 5.0/RTOG criteria.

SECONDARY OUTCOMES:
Local Regional Relapse-Free Survival (LRRFS) | 5 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Distant Metastasis-Free Survival (DMFS) | 5 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Progress-Free Survival (PFS) | 5 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.
The proportion of patients with treatment related complications | 5 years
  The proportion of patients with treatment related complications according to NCI-CTC5.0 criteria and RTOG criteria.
Objective response rate (ORR) | 3 months
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to treatment. (according to tumor imaging examinations 3 months after the end of treatment/supplementary treatment)
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 5 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 5 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China